CLINICAL TRIAL: NCT02720601
Title: A Phase II Trial of Combination Irinotecan and Capecitabine as Second-Line Treatment for Patients With Locally Advanced/Metastatic Biliary Tract Cancers Who Progressed or Intolerant to Front-Line Gemcitabine and Platinum Combination
Brief Title: Irinotecan and Capecitabine as Second-line Treatment for Advanced/Metastatic Biliary Tract Cancers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never submitted to the IRB & never opened. PI is leaving institution.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1417
Record Dates: First submitted 2016-03-23; First posted 2016-03-28 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Biliary Tract Cancer
Keywords: irinotecan; capecitabine; gemcitabine; biliary tract cancer; gallbladder cancer; second-line
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms | interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan & Capecitabine (Experimental): Irinotecan at 120 mg/m2 intravenously every three weeks + Capecitabine at 1500 mg/m2/day orally twice per day for a total of 14 days.
  The treatment cycle is once every 21 days.
  Interventions: Drug: Irinotecan & Capecitabine

INTERVENTIONS:
Drug: Irinotecan & Capecitabine — Irinotecan will be administered at infusion room over 60 minutes. Capecitabine will be administered by the patients at home. Unless there is early progression of disease, at least two courses will be administered to each patient. Repeated courses may be given to the patients who benefit from the treatment (either complete or partial remission, or stabilization of disease)
  Other Names: Irinotecan = Camptosar, Campto, or CPT-11 (Camptothecin-11); Capecitabine = Xeloda

SUMMARY:
Biliary tract cancers that progress after first line treatment can be difficult to treat. There is a great need for an effective, tolerable, easy to administer second-line regimen. Previous early phase studies demonstrated that the combination of two chemotherapy drugs, irinotecan and capecitabine had activity in this setting. The goal of this study is to determine whether this drug combination, as a second-line treatment, can improve progression free survival in patients with biliary tract cancers.

DETAILED DESCRIPTION:
The current front-line treatment regimen using gemcitabine in combination with cisplatin has a significant survival benefit (11.7 versus 8.1 months, P < 0.001) in patients with biliary tract cancer when compare to single agent gemcitabine. However, there is urgent need for effective second-line regimens with minimal toxicity.

Capecitabine (Xeloda) is an oral pro-drug of 5-fluorouracil (5-FU). The conversion to active drug is dependent on thymidine phosphorylase, which is expressed at a higher level in tumor cells than in normal tissue. There are no reports on prospective clinical trials using capecitabine in cholangiocarcinoma. However, case reports of successful stabilization of disease with single agent capecitabine are available. Since 5-FU has been the main chemotherapy agent for biliary tract cancer for more than 40 years, it is reasonable to presume that the overall effectiveness of capecitabine will be very similar to infusional 5-FU.

Several clinical trials have shown that irinotecan can be a good agent for cholangiocarcinoma. Of the five patients that had a partial response in one phase I trial of the combination of irinotecan and docetaxel in advanced solid tumors, one had cholangiocarcinoma. Two of the 11 patients that had a partial response from another phase I trial using a combination of irinotecan, oxaliplatin and 5-FU in advanced tumors had cholangiocarcinoma. A case report indicated that single agent irinotecan given at a low weekly dose could produce a long-lasting response in metastatic cholangiocarcinoma.

Based on the above data, our experience, and other early phase studies of this combination, this phase II trial was proposed to determine the progression free survival, response rate, overall survival, and toxicity in biliary tract cancer patients who are administered irinotecan and capecitabine as a second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Histological proven un-resectable or metastatic biliary tract cancer (gallbladder cancer included) with radiologic progression after initial gemcitabine plus platinum (cisplatin, carboplatin or oxaliplatin) regimen
* Computerized tomography (CT) or magnetic resonance imaging (MRI) with measurable lesions no more than 28 days prior to enrollment. Lesions should be at least 1.5 cm in longest dimension.
* Patients with evaluable only disease, effusion, needs to have cytology proven malignant cells present in the effusion.
* Patients who cannot tolerate or developed allergic reaction to either gemcitabine or platinum compounds, even without radiographic progression will be eligible.
* Patients must have a life expectancy of at least 12 weeks
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
* Patients must be able to understand and sign informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of ≥ 1,500 cells/mm3 and platelet count ≥ 60,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin ≤ 4.0 mg/dl, could be ≤ 10 mg/dl if a functional biliary drain is placed within three days of enrollment and documented declining total bilirubin level, and adequate renal function as defined by a serum creatinine ≤ 1.5 X upper limit of normal.
* Patients with concurrent basal cell carcinoma and/or squamous cell carcinoma of skin are eligible.
* Patients with other malignancies require having at least 5 year disease-free interval before enrollment
* Patients who were treated with either irinotecan and/or capecitabine for cancers other than biliary tract cancer are eligible as long as treatment-free interval is greater than 3 years.

Exclusion Criteria:

* Patients with symptomatic central nervous system (CNS) metastases are excluded. Need to demonstrate stable CNS metastases for at least 3 months
* Pregnant women and nursing mothers are not eligible.
* Patients of child bearing potential must agree to use adequate contraception
* No heart attack within 6 months of enrollment
* No stroke (embolic and hemorrhage) within 6 months of enrollment.
* No New York Heart Association Class III/IV congestive heart failure (CHF).
* Severe chronic obstructive pulmonary disease (COPD) requires ≥ 2 L (Liters) /minute of oxygen.
* Known history of allergic reaction to irinotecan and/or capecitabine.
* Known history of 5-fluorouracil (5-FU) or capecitabine induced cardiac toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months from the time of initiating treatment
  The time from initiation of treatment to disease progression or death by any cause. Progression is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1). Progressive disease (PD) for target lesions: >= 20% increase in the sum of diameters of the target lesions taking as reference the smallest sum on study, and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered . PD for non-target lesions is defined as unequivocal appearance of one or more new malignant lesions or unequivocal progression of existing non-target lesions.The Kaplan-Meier method will be used to calculate the proportion of subjects who are progression-free at 6 months along with its 95% confidence interval. Subjects lost to follow-up or who withdraw from the study for any reason will be censored at their last date of contact

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 6 months after initiating treatment
  Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1). Complete response (CR): Disappearance of all evidence of target and non-target lesions. Partial response (PR): >= 30% reduction from baseline in the sum of the longest diameter of all lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks after initial assessment. Best overall response is the best response recorded from the start of treatment until disease progression/recurrence. (For definition of progression, see Outcome Measure 1). Overall response rate will be reported as the sum of the percentages of patients achieving CR and PR.
Overall Survival (OS) | 36 months from enrollment
  The time from study enrollment to death by any cause. Subjects who withdraw from the study for any reason or are lost to follow-up will be censored at their last date of contact. The Kaplan-Meier method will be used to calculate the median OS and 95% confidence interval
Toxicity | Up to 30 days after last on-study treatment
  Toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE), ver. 4.0. Adverse events of grade 3 or higher will be reported as percentages of patients affected. If subjects experience the same toxicity more than once, the subjects' highest grade toxicity will be used for summaries.

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, MD, Principal Investigator — University of New Mexico
Locations (1):
- Universtiy of New Mexico - Cancer Center, Albuquerque, New Mexico, United States